CLINICAL TRIAL: NCT07097480
Title: Virus Transmission to People Recently Bitten or With a History of Monkey Bites "SIMVIR"
Brief Title: Virus Transmission to People Recently Bitten or With a History of Monkey Bites "SIMVIR
Acronym: SIMVIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-113
Record Dates: First submitted 2025-07-25; First posted 2025-07-31 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-07

CONDITIONS: Bites Monkey
Keywords: Antirabies; Virus; Bite; Infection
MeSH Terms: conditions — Virus Diseases; Bites and Stings; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adults recently bitten by a non-human primate (Other): Adults recently bitten by a non-human primate and consulting at the Institut Pasteur medical center for prophylaxis as part of their care.
  Interventions: Procedure: Blood samples collection; Procedure: Saliva samples collection
- Adults with a history of bites (Other): Adults with a history of bites from a non-human primate who are consulting at the Institut Pasteur medical center as part of their routine care.
  Interventions: Procedure: Blood samples collection; Procedure: Saliva samples collection

INTERVENTIONS:
Procedure: Blood samples collection — Blood samples of 40 ml will be taken.
Procedure: Saliva samples collection — Saliva samples will be collected

SUMMARY:
Nonhuman primates (NHPs) constitute an important reservoir of infectious agents, some of which have emerged in human populations as deadly pathogens. Human exposure to the biological fluids of NHPs - particularly through bites - can result in the transmission of several viruses. Only the rabies virus is currently targeted by post-exposure prophylaxis following an injury caused by an NHP.

The objective of the study is to investigate the prevalence of STLV-1 and SFV infections following a nonhuman primate bite.

DETAILED DESCRIPTION:
Nonhuman primates (NHPs) constitute an important reservoir of infectious agents, some of which have emerged in human populations as deadly pathogens. Human exposure to the biological fluids of NHPs - particularly through bites - can result in the transmission of several viruses. Only the rabies virus is currently targeted by post-exposure prophylaxis following an injury caused by an NHP.

Compared to other individuals exposed to nonhuman primates (NHPs), travelers have two unique characteristics. First, they are typically exposed only once to simian infectious agents, in contrast to the repeated exposure experienced by other at-risk groups. If exposure results in an infection event, travelers may spread these infectious agents to geographic areas where they do not normally circulate.

To address the following main objective: to study the prevalence of STLV-1 and SFV infections following a nonhuman primate bite. The study plans to include subjects who have been recently bitten as well as those with a history of nonhuman primate bites. Blood and saliva samples will be collected from the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Bite inflicted by an HNP (WHO category 3 level)
* Written informed consent
* Affiliation with a social security scheme (excluding State Medical Aid

Specific criteria for genetic analyses:

* Participant has checked the boxes for participation in the genetic component.

Exclusion Criteria:

* Patient presenting only with scratches inflicted by a PNH
* Medical management incompatible with the objectives of the study
* Patient who, in the doctor's opinion, is unlikely to comply with the study protocol
* Health conditions are incompatible with the sample collection required by the study
* Patient under legal protection (guardianship or trusteeship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Study the prevalence of STLV-1 and SFV infections following an NHP bite. | 17 months
  Detection of specific antibodies and viral DNA against both viruses in blood.

SECONDARY OUTCOMES:
Identify risk and demographic factors associated with STLV-1 and SFV infection. | 17 months
  The study of associations between STLV-1 and SFV infection and demographic characteristics (age, sex) and those linked to the HNP bite (severity of injury, HNP species) will be analyzed by Fisher's exact test and the Mann-Withney test.

OTHER OUTCOMES:
Determine the kinetics of appearance of viral markers (viral DNA and antibodies) for each virus | 17 months
  Measurement of viral markers (SFV RNA and DNA, STLV-1 DNA, virus-specific IgM and IgG) in blood and saliva.
Characterize detected STLV-1 and SFV viral strains | 17 months
  Determination of complete viral sequences and integration sites in the human genome.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick HOCHEDEZ, Dr, Principal Investigator — Institut Pasteur Medical Center
Locations (1):
- Institut Pasteur Medical Center, Paris, France